CLINICAL TRIAL: NCT00757978
Title: Phase 4 Memantine as Adjunctive Therapy for Schizophrenia Negative Symptoms in Patients Using Clozapine. A Randomized, Double-Blind, Placebo Controled Study
Brief Title: Memantine as Adjunctive Therapy for Schizophrenia Negative Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: FIPE, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-406; FIPE-HCPA 05-406
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; negative symptoms; clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Memantine; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Clozapine plus placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): Clozapine plus memantine
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — memantine 10mg twice a day
  Other Names: Ebixa
  Arms: 2
Drug: placebo — 1 capsule of placebo twice a day
  Other Names: Starch
  Arms: 1

SUMMARY:
Memantine as an add-on therapy to clozapine may improve schizophrenia negative symptoms and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Under clozapine with negative symptoms

Exclusion Criteria:

* Pregnancy
* Lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Score in Brief Psychiatric Raring Scale | baseline, 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa S Gama, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Lucena D, Fernandes BS, Berk M, Dodd S, Medeiros DW, Pedrini M, Kunz M, Gomes FA, Giglio LF, Lobato MI, Belmonte-de-Abreu PS, Gama CS. Improvement of negative and positive symptoms in treatment-refractory schizophrenia: a double-blind, randomized, placebo-controlled trial with memantine as add-on therapy to clozapine. J Clin Psychiatry. 2009 Oct;70(10):1416-23. doi: 10.4088/JCP.08m04935gry. PMID 19906345